CLINICAL TRIAL: NCT00132392
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Analgesic Efficacy, Safety and Tolerability of ALGRX 4975 in Subjects After Total Knee Arthroplasty
Brief Title: ALGRX 4975 After Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoRx Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4975-2-010-1
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2005-08

CONDITIONS: Arthroplasty, Replacement, Knee; Knee Injuries
Keywords: Arthroplasty; Total knee arthroplasty; Capsaicin; Pain; Analgesia
MeSH Terms: conditions — Knee Injuries; Pain; Agnosia

INTERVENTIONS:
Drug: ALGRX 4975

SUMMARY:
ALGRX 4975 or placebo will be dripped onto the cut muscles and soft tissues before the end of surgery for total replacement of the knee.

Each subject will undergo a screening visit; a hospitalization, during which total replacement of the knee will be performed; and follow-up visits at 2, 6, and 12 weeks after surgery. In addition, once discharged, subjects will be contacted by telephone daily up to Day 14. Subjects will complete pain and medication diaries during the first 2 weeks following surgery and will return these diaries at the 2 week visit.

Starting on the afternoon of Day 0 (the day of surgery), pain on active range of motion (ROM) of the operated knee will be measured each morning at 8 AM ± 2 hours and each afternoon at 3 PM ± 3 hours. In addition, if the subject ambulates, pain with ambulation will be measured during the first ambulation in the morning and during the first ambulation after noon. Subjects will complete the Brief Pain Inventory - Short Form (BPI-SF) preoperatively, and at the 2, 6, and 12 week visits. Subjects will be questioned regarding the use of assistive devices (cane, walker, wheelchair, bedside commode, or other assistive devices) at screening, at discharge, and at the 2, 6, and 12 week visits. The active ROM on flexion of the knee, measured using a goniometer, will be recorded at screening and at the 2 week visit. Sensory mapping of the knee will be performed at screening and at the 12 week visit.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, study conducted in subjects undergoing unilateral TKA. Subjects will undergo a screening visit up to 28 days prior to surgery. A sufficient number of subjects will be enrolled to obtain at least 40 evaluable subjects. Upon enrollment, subjects will be randomized in a 1:1 ratio of ALGRX 4975 to placebo. Subjects will receive a femoral nerve block prior to induction of general anesthesia. Subjects will undergo total knee arthroplasty (TKA) under general anesthesia. Prior to closure of the surgical wound, a single dose of ALGRX 4975 5 mg in 60 mL or placebo will be instilled (dripped by syringe over approximately 1 minute) into the wound onto the cut muscles and soft tissues and allowed to dwell for 5 minutes. The Investigator will then inject bupivacaine 0.25% up to 40 mL into the area of the wound and cut muscles and close the wound by usual surgical procedures. Postoperative pain will be managed by morphine sulfate administered intravenously by patient controlled analgesia (PCA). Following discontinuation of the PCA pump, subjects will be provided with hydrocodone 7.5 mg/acetaminophen 500 mg for postoperative pain.

Each subject will undergo a screening visit; a hospitalization, during which TKA will be performed; and follow-up visits at 2, 6, and 12 weeks after surgery. Subjects will receive twice daily examinations while hospitalized for the TKA procedure. In addition, once discharged, subjects will be contacted by telephone daily up to Day 14, to remind them to complete pain and medication diaries, and then again at 4 weeks after surgery for follow-up. Subjects will complete pain and medication diaries during the first 2 weeks following surgery and will return these diaries at the 2 week visit.

Starting on the afternoon of Day 0 (the day of surgery), pain on active range of motion (ROM) of the operated knee will be measured using an 11 point numerical rating scale (NRS) each morning at 8 AM ± 2 hours and each afternoon at 3 PM ± 3 hours, not within one hour after physical therapy. In addition, if the subject ambulates, pain with ambulation will be measured during the first ambulation in the morning and during the first ambulation after noon. Subjects will complete the Brief Pain Inventory - Short Form (BPI-SF) preoperatively, and at the 2, 6, and 12 week visits. Subjects will be questioned regarding the use of assistive devices (cane, walker, wheelchair, bedside commode, or other assistive devices) at screening, at discharge, and at the 2, 6, and 12 week visits. The active ROM on flexion of the knee, measured using a goniometer, will be recorded at screening and at the 2 week visit. Sensory mapping of the knee will be performed at screening and at the 12 week visit.

ELIGIBILITY:
Inclusion Criteria:

* The subject (male or female) is aged 35 - 80 years. Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to administration of study drug; must be nonlactating; and must be willing to use adequate and reliable contraception throughout the study.
* The subject is planned to undergo unilateral TKA.
* The subject is willing and able to understand the study procedures and the use of pain scales, and to communicate meaningfully with the study personnel.
* The subject is in good health and capable of undergoing TKA.
* The subject has signed the Informed Consent approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* The subject has a laboratory test value outside the accepted range unless approved by the Sponsor.
* The subject is currently taking or has taken a chronic opioid (more than 30 consecutive days of daily use) for pain other than knee pain in the past two years.
* The use of capsaicin, opioids, bupivacaine, ropivacaine, muscle relaxants, or acetaminophen is contraindicated in this subject (e.g., significant history of allergic reactions or intolerance to these or related substances).
* The use of general anesthesia is contraindicated in this subject.
* The subject is taking central nervous system (CNS) active drugs such as benzodiazepines, tricyclic antidepressants, or selective serotonin reuptake inhibitors (SSRIs) for pain. These drugs are permitted for non-pain indications if the dose has been stable for at least 30 days. The use of non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen is permitted if stable over at least 30 days. The use of lorazepam and other sleep medications is permitted. Administration of ketorolac tromethamine (Toradol®) is permitted preoperatively, intraoperatively, and postoperatively no later than 8 PM on the day of surgery.
* The subject has a medical condition that, in the Investigator's opinion, could adversely impact the subject's participation or safety; conduct of the study; or interfere with the pain assessments, including fracture or active infection.
* The subject has diabetes mellitus and HbA1C > 9.5 or a history of prolonged uncontrolled diabetes.
* The subject has another painful physical condition that, in the opinion of the Investigator, may confound the assessments of postoperative pain or rehabilitation. The subject has a history of or current neuropathic pain condition.
* The subject is planned to undergo bilateral TKA.
* The subject has had arthroplasty (partial or total) of the index knee.
* The subject has a history of drug, prescription medicine or alcohol abuse within the past 2 years.
* The subject is taking an antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days
* The subject is taking any of the following medications: digoxin; all antiarrhythmics except beta-blockers; warfarin; theophylline preparations; aminoglycosides; anticonvulsants except benzodiazepines; and lithium.
* The subject has taken an investigational product within 3 months prior to the first dose of study drug (Visit 2), or is scheduled to receive an investigational product other than ALGRX 4975, while participating in the study.
* The subject has a known bleeding disorder or is taking agents affecting coagulation. Low dose aspirin is allowed as cardiac prophylaxis; NSAIDs, if stable for at least 30 days, are permitted; and deep venous thrombosis prophylaxis, of the surgeon's choice, is permitted postoperatively.
* The subject has previously participated in a clinical study with ALGRX 4975.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-07; Study Completion 2005-12

PRIMARY OUTCOMES:
The daily average of the numerical rating scale (NRS) for pain with active range of motion of the operated knee at 8 AM ± 2 hours and at 3 PM ± 3 hours on Day 1, on Day 2, and on Days 1 through 2

SECONDARY OUTCOMES:
The daily average of the numerical rating for pain with active range of motion of the operated knee at 8 AM ± 2 hours and at 3 PM ± 3 hours on Days 3 through 14, and Days 1 through 14
The daily average of the numerical rating for pain during first ambulation in the morning and first ambulation after noon on Day 1, Day 2, Days 1 through 14, and Days 3 through 14
Morphine sulfate that the subject self-administers for postoperative pain for each 12 hour period postoperatively starting at 8 AM on the day following surgery
Time to first dose of supplemental pain medication (hydrocodone 7.5 mg/acetaminophen 500 mg) after self-administration of morphine sulfate is discontinued
Number of tablets of hydrocodone 7.5 mg/acetaminophen 500 mg used during the first two postoperative weeks after total knee arthroplasty (TKA)
The average quantity of hydrocodone 7.5 mg/acetaminophen 500 mg used during the first two postoperative weeks after surgery
Pain and pain interference with activities at 2, 6, and 12 weeks using the Brief Pain Inventory-Short Form (BPI-SF)
Effect of ALGRX 4975 on the use of assistive devices (cane, walker, wheelchair, bedside commode, or other assistive devices) at discharge, 2, 6, and 12 weeks
Effect of ALGRX 4975 on active flexion range of motion of the operated knee, measured using a goniometer, at the 2 week postoperative visit

CONTACTS AND LOCATIONS:
Locations (1):
- Capstone Clinical Trials, Inc., Birmingham, Alabama, United States